CLINICAL TRIAL: NCT04719234
Title: Comparison of Lung Ultrasonography Findings With Chest Computerized Tomography Results in Corona virüs (COVID-19) Pneumonia
Brief Title: Lung Ultrasonography in COVID-19 Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Korgün Ökmen, Principal Investigator ,Assoc. PhD. M.D., Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011-KAEK-25 2020/5-21
Record Dates: First submitted 2021-01-20; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Lung Ultrasound; Pneumonia; Covid19
MeSH Terms: conditions — Pneumonia; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- lung ultrasound (Other): lung ultrasonography protocol will be applied.
  Interventions: Device: lung ultrasonography

INTERVENTIONS:
Device: lung ultrasonography — Application of 12 zone lung ultrasonography protocol using the konvex ultrasound probe (2-6 MHz)

SUMMARY:
Lung ultrasonography has been used for diagnosis and treatment in many departments including intensive care before the pandemic. The gold standard method for the diagnosis of pneumonia is still chest tomography. Ultrasonography, which has advantages over tomography, has also been tried to be used in covid 19 pneumonia.

DETAILED DESCRIPTION:
In this study, it was aimed to investigate the efficiency of lung ultrasonography in diagnosis of covid 19 pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* 18 and 85 years old
* Hospitalized in intensive care unit
* PCR tested
* Thoracic CT applied

Exclusion Criteria:

* Previous lung and thoracic wall surgery
* Anatomically with thoracic wall disorder
* Patients who did not consent to participate in the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Relationship between Thoracic CT imaging results and LUS results | 6 hours
  Lung ultrasonography will be performed within 6 hours of the Thoracic CT.

SECONDARY OUTCOMES:
Characteristics of lesions | 6 hours
  İdentifying the characteristics of the abnormal findings detected in Thoracic CT and LUS

OTHER OUTCOMES:
the relation of the lesions with the pleura | 6 hours
  the relation of the lesions with the pleura, and their distance to the pleura.

CONTACTS AND LOCATIONS:
Overall Officials: Korgün Ökmen, Assoc. PhD., Principal Investigator — Sağlık Bilimleri Üniversitesi Bursa Yüksek İhtisas Eğitim Ve Araştırma Hastanesi; Durdu Kahraman Yıldız, M.D, Study Chair — Sağlık Bilimleri Üniversitesi Bursa Yüksek İhtisas Eğitim Ve Araştırma Hastanesi; Emel Tatar Soyaslan, M.D, Study Chair — Sağlık Bilimleri Üniversitesi Bursa Yüksek İhtisas Eğitim Ve Araştırma Hastanesi
Locations (1):
- University of Health Sciences, Bursa Yuksek Ihtisas Training and Research Hospital, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Okmen K, Yildiz DK, Soyaslan E. Comparison of lung ultrasonography findings with chest computed tomography results in coronavirus (COVID-19) pneumonia. J Med Ultrason (2001). 2021 Apr;48(2):245-252. doi: 10.1007/s10396-021-01081-7. Epub 2021 Feb 26. PMID 33638057